CLINICAL TRIAL: NCT05462821
Title: Randomized Trial of Full-Time Occlusion Therapy for Intermittent Exotropia in Children
Brief Title: Full-Time Occlusion Therapy for Intermittent Exotropia in Children
Acronym: IXT7
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH); Pediatric Eye Disease Investigator Group (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IXT7; 2U10EY011751 (NIH)
Record Dates: First submitted 2022-07-14; First posted 2022-07-18 (Actual); Results first posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Intermittent Exotropia
Keywords: IXT; intermittent exotropia; occlusion therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Observation Group (No Intervention): Participants randomized to observation alone will not be allowed to receive any other treatment for IXT, except refractive correction, for 3 months.
- Full Time Patching (Experimental): Participants randomized to the full-time patching group will patch full-time (all waking hours) for 3 months up until the day before the 3-month primary outcome visit. Daily alternate patching will be prescribed (right eye on even days, left eye on odd days). No other treatment for IXT will be used, except for refractive correction.
  Interventions: Device: Eye Patch

INTERVENTIONS:
Device: Eye Patch — adhesive patch to cover eye
  Arms: Full Time Patching

SUMMARY:
Determine whether full-time patching is more effective than observation for improving distance control of IXT after 3 months of treatment (on-treatment outcome).

DETAILED DESCRIPTION:
Understanding the effectiveness of intensive patching has important implications for managing children with IXT. If full-time patching is associated with improvement in distance control vs an observation group, then future studies can be conducted to evaluate different durations of full-time patching treatment, whether the effect is maintained off-treatment, and how full-time patching compares to other treatment strategies.

The purpose of this study is to determine whether full-time patching is more effective than observation for improving distance control of IXT after 3 months of treatment (on-treatment outcome).

ELIGIBILITY:
Inclusion Criteria:

Children under the care of a pediatric optometrist or pediatric ophthalmologist will be eligible for the study if they meet all the following criteria:

1. Age 3 to < 9 years
2. IXT meeting all of the following criteria:

   * Intermittent or constant XT at distance (mean distance control 2.0 or more) with at least 1 control measure of 3, 4 or 5 (i.e., indicating spontaneous tropia)
   * Either IXT, exophoria, or orthophoria at near (cannot have control score of 5 on all 3 near assessments)
   * Distance exodeviation between 15∆ and 50∆ by PACT
   * Near exodeviation between 0∆ and 50∆ by PACT
   * Near exodeviation does not exceed distance by more than 10∆ by PACT (convergence insufficiency-type IXT excluded)
3. Age-normal visual acuity in both eyes:

   * 3 years: 20/50 or better (>=63 letters)
   * 4 years: 20/40 or better (>=68 letters)
   * 5-6 years: 20/32 or better (>=73 letters)
   * 7-<9 years: 20/25 or better (>=78 letters)
4. Interocular difference in distance VA of 2 logMAR lines or less (10 letters or less on E-ETDRS for patients ≥7 years old). Testing by ATS HOTV for participants 3 to < 7 years old and by E-ETDRS for participants ≥7 years old.
5. Cycloplegic refraction within the last 7 months.
6. Refractive error between -6.00 D SE and +2.00 D SE (inclusive) based on a cycloplegic refraction within 7 months
7. Participants with refractive error meeting any of the following based on a cycloplegic refraction within 6 months must be wearing spectacles for at least 2 weeks:

   * Myopia > -0.50 D spherical equivalent (SE) in either eye
   * Anisometropia > 1.00 D SE
   * Astigmatism in either eye > 1.00 D
8. Any refractive correction worn at enrollment (required or not) must meet the following guidelines based on a cycloplegic refraction within 7 months:

   * Anisometropia SE must be within 0.50 D of the full anisometropic difference correction
   * Astigmatism must be corrected within 0.50 D
   * Axis must be within ±10 degrees if cylinder power is ≤1.00 D and within ±5 degrees if cylinder power is >1.00 D.
   * For hyperopia, the spherical component can be reduced at investigator discretion provided the reduction is symmetrical and does not meet the definition of deliberate overminus (see below).
   * For myopia, the intent is to fully correct, but the spherical component can be undercorrected at investigator discretion provided the reduction is symmetrical and results in no more than -0.50 D SE residual (i.e., uncorrected) myopia. Deliberate overminus is not allowed.
   * Deliberate overminus is defined for this protocol as any refractive correction prescribed to yield lenses that are overminused by more than -0.50D SE than cycloplegic refraction SE

     * Less than the full cycloplegic hyperopic correction (i.e., prescribing reduced plus) is not considered the same as overminusing for this protocol (because most patients without IXT but with hyperopic SE refractions up to +2.00 D SE would not typically be prescribed a refractive correction.)
   * For refractive errors with an emmetropic or myopic SE, the intent is to fully correct, but the spherical component can be undercorrected at investigator discretion provided the reduction is symmetrical and results in no more than -0.50 D SE residual (i.e., uncorrected) myopia. Prescribing a correction that yields more than 0.50 D more minus SE than the cycloplegic refraction SE is considered deliberate overminus and is not allowed.
   * Note that the refractive correction guidelines and the requirement to wear refractive correction for at least 2 weeks apply not only to participants who require refractive correction under the above criteria but also to any other participant who is wearing refractive correction.
9. Gestational age > 30 weeks
10. Birth weight > 1500 grams
11. Patient and/or parent understands protocol, is willing to enroll, and is willing to accept that other (i.e., nonrandomized) treatment for IXT will not be offered by the investigator for 3 months
12. Parent has phone and is willing to be contacted by Jaeb Center staff
13. Relocation outside of area of an active PEDIG site within 3 months not anticipated

Exclusion Criteria:

Individuals meeting any of the following criteria at baseline will be excluded from study participation:

1. Prior strabismus, intraocular, or refractive surgery (including BOTOX injection)
2. Prior nonsurgical treatment for IXT (e.g., patching, vergence therapy, vision therapy/orthoptics, base-in prism, or deliberate overminus (more than 1.00 D) spectacles of >1week duration within the past year
3. Previous amblyopia treatment other than refractive correction
4. Diplopia more than 2 times per day by parental assessment
5. Paretic or restrictive strabismus
6. Craniofacial malformations affecting the orbits
7. Ocular disorders which would reduce VA (except refractive error)
8. Severe developmental delay that would interfere with treatment or evaluation (in the opinion of the investigator). Participants with mild speech delay or reading and/or learning disabilities or ADHD are not excluded.
9. Neurological anomaly that could affect ocular motility (e.g., cerebral palsy, Down syndrome)
10. Immediate family member (child or sibling) of any investigative site personnel directly affiliated with this study.
11. Known allergy to adhesive patches.
12. Known allergy to silicone.

Ages: 3 Years to 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 73 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-05-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen P Christiansen, MD, Study Chair — Boston Children's Hospital; Erin C Jenewein, OD, Study Chair — Salus University
Locations (25):
- United States (25):
  - UAB Pediatric Eye Care; Birmingham Health Care, Birmingham, Alabama
  - Arkansas Childrens, Little Rock, Arkansas
  - Univ. of California- Berkeley, Berkeley, California
  - Southern California College of Optometry, Fullerton, California
  - Univ of California, Irvine- Gavin Herbert Eye Institute, Irvine, California
  - Loma Linda University Health Care, Dept. of Ophthalmology, Loma Linda, California
  - Stanford University, Palo Alto, California
  - Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Progressive Eye Care, Lisle, Illinois
  - Indiana School of Optometry, Bloomington, Indiana
  - Wilmer Eye Institute, Baltimore, Maryland
  - Boston Medical Center, Boston, Massachusetts
  - Boston Children's Hospital Waltham, Boston, Massachusetts
  - Michigan College of Optometry at Ferris State Univ, Big Rapids, Michigan
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - State University of New York, College of Optometry, New York, New York
  - Duke University Eye Center, Durham, North Carolina
  - Ohio State University College of Optometry, Columbus, Ohio
  - Eye Care Associates, Inc., Poland, Ohio
  - Casey Eye Institute, Portland, Oregon
  - Salus University/Pennsylvania College of Optometry, Philadelphia, Pennsylvania
  - Southern College of Optometry, Memphis, Tennessee
  - Virginia Pediatric Eye Center, Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: Yes
In accordance with the NIH data sharing policy, a de-identified database is placed in the public domain on the PEDIG public website after the completion of each protocol and publication of the primary manuscript.
Supporting Information: Study Protocol
Time Frame: Data will be made available after publication of each primary manuscript
Access Criteria: Users accessing the data must enter an email address.
URL: http://pedig.jaeb.org/

REFERENCES:
- [Background] Hatt SR, Leske DA, Holmes JM, Henderson RJ, Chandler DL, Morrison DG, Summers AI, Cotter SA. Testing depth of suppression in childhood intermittent exotropia. J AAPOS. 2022 Feb;26(1):36-38.e1. doi: 10.1016/j.jaapos.2021.08.303. Epub 2021 Nov 16. PMID 34793970

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Observation Group | Full Time Patching
Started | 37 | 36
Completed | 35 | 33
Not Completed | 2 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Observation Group | Full Time Patching | Total
Number analyzed (Participants) | 37 | 36 | 73
Age, Customized [Count of Participants; unit: Participants]
  3 years old | 5 | 5 | 10
  4 years old | 8 | 12 | 20
  5 years old | 8 | 5 | 13
  6 years old | 6 | 5 | 11
  7 years old | 8 | 6 | 14
  8 years old | 2 | 3 | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 16 | 12 | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 11 | 11 | 22
  Not Hispanic or Latino | 26 | 25 | 51
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 1 | 3
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 8 | 6 | 14
  White | 19 | 17 | 36
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 3 | 5 | 8
Prior Non-Surgical Treatments for IXT [Count of Participants; unit: Participants]
  Overminus > 1 year prior to enrollment | 1 | 1 | 2
  Patching > 1 year prior to enrollment | 1 | 1 | 2
  Prism > 1 year prior to enrollment | 1 | 0 | 1
  Pencil Push-Ups within 1 year prior to enrollment (patient ineligible) | 1 | 0 | 1
  None | 33 | 34 | 67
Neurological Anomaly That Could Affect Ocular Motility? [Count of Participants; unit: Participants]
  Yes (patient ineligible) | 1 | 0 | 1
  No | 36 | 36 | 72
Spectacle Status [Count of Participants; unit: Participants]
  Not wearing spectacles | 26 | 26 | 52
  Wearing spectacles at least two weeks | 11 | 10 | 21
Stereoacuity at near, arcseconds (log10 arcseconds) [Count of Participants; unit: Participants] — Randot® Preschool Stereoacuity test (Stereo Optical Co., Inc., Chicago, IL). For analysis, stereoacuity was converted from seconds of arc scores to log10 arcsec values. Children with no detectable (nil) stereoacuity were assigned the value of 1600 arcsec (3.20 log10 arcsec).
  Participants
    40 (1.60) | 5 | 8 | 13
    60 (1.78) | 12 | 9 | 21
    100 (2.00) | 6 | 6 | 12
    200 (2.30) | 5 | 3 | 8
    400 (2.60) | 4 | 3 | 7
    800 (2.90) | 1 | 3 | 4
    Nil (3.20) | 2 | 2 | 4
    Unable to Complete pretest | 2 | 2 | 4
Participant Baseline Suppression Scores [Count of Participants; unit: Participants] — The Office Suppression Test standardizes the grading of suppression in intermittent exotropia when manifest (induced if not present). A single 20/50 optotype is viewed at 6 meters in normal room lighting; if 2 letters are seen, suppression is "negligible" (scored 0). If only 1 letter is seen a 6-meter light is viewed with a red filter over the fixing eye in normal lighting. If 2 lights are seen (1 white, 1 red), suppression is graded "mild," (scored 1). If only 1 light is seen, room lights are dimmed; 2 lights is graded "moderate" (scored 2) whereas 1 light is graded "dense" (scored 3).
  Participants
    Negligible (0) | 9 | 4 | 13
    Mild (1) | 5 | 5 | 10
    Moderate (2) | 7 | 9 | 16
    Dense (3) | 11 | 12 | 23
    Missing (children were unable to understand the test and/or gave unreliable responses) | 5 | 6 | 11
Interocular Difference in Visual Acuity (logMAR lines) [Count of Participants; unit: Participants]
  Within one line (0 to <1) | 24 | 21 | 45
  One line (1 to <2) | 10 | 11 | 21
  Two lines (=2) | 3 | 4 | 7
Average OD/OS Visual Acuity Snellen Equivalent (logMAR) [Count of Participants; unit: Participants]
  20/12 (-0.2) | 1 | 1 | 2
  20/16 (-0.1) | 8 | 10 | 18
  20/20 (0.0) | 10 | 8 | 18
  20/25 (0.1) | 12 | 8 | 20
  20/32 (0.2) | 3 | 5 | 8
  20/40 (0.3) | 2 | 4 | 6
  20/50 (0.4) | 1 | 0 | 1
Average OD/OS Spherical Equivalent Refractive Error, D [Count of Participants; unit: Participants]
  -6.00 to <-0.50 D | 4 | 5 | 9
  -0.50 to <0.50 D | 13 | 13 | 26
  0.50 to <2.00D | 20 | 18 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Change in Mean Distance Control Scores at 3 Months
Description: To determine if participants with IXT undergoing full-time patching have more improvement in mean distance control between baseline and 3 months than participants being observed without treatment.
  The Office Control Score provides a rating of exodeviation control on a 0 to 5 scale, in subjects with intermittent exotropia. Scores 3 to 5 reflect the proportion of time a spontaneous manifest exotropia is present during 30 seconds of observation (<50% score 3; >50% score 4; 100% score 5). If no spontaneous manifest exotropia is observed, scores 0 to 2 reflect the longest time to regain fusion after three, 10-second dissociations (>5 seconds score 2; 1-5 seconds score 1; <1 second score 0).
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Observation Group | Full Time Patching
Number analyzed (Participants) | 35 | 33
Participants
  2 to <3 | 1 | 0
  1 to <2 | 4 | 4
  0 to <1 | 13 | 8
  -1 to <0 | 7 | 3
  -2 to <-1 | 8 | 9
  -3 to <-2 | 1 | 7
  -4 to <-3 | 1 | 2

ADVERSE EVENTS:
Time Frame: Adverse events were monitored/assessed from the participant's perspective between randomization and completion of their 3 month primary outcome visit.
Description: No adverse events are anticipated as a result of alternating full-time patching or as a result of observation. No surgical procedures are part of the protocol and no treatments are being prescribed that are not part of usual care. Symptom survey data have been reported as outcomes by treatment group.
Arm/Group | Observation Group | Full Time Patching
All-Cause Mortality (participants affected / at risk) | 0/35 | 0/33
Serious Adverse Events (participants affected / at risk) | 0/35 | 0/33
Other Adverse Events (participants affected / at risk) | 0/35 | 0/33

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2022-04-19): https://cdn.clinicaltrials.gov/large-docs/21/NCT05462821/Prot_000.pdf
  • Statistical Analysis Plan (2025-05-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT05462821/SAP_002.pdf
  • Informed Consent Form (2022-06-30): https://cdn.clinicaltrials.gov/large-docs/21/NCT05462821/ICF_001.pdf